CLINICAL TRIAL: NCT07403188
Title: A Long-Term Follow-Up Study for Participants Previously Treated With KYV-101
Acronym: KYSA-4
Status: Recruiting | Type: Observational
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: KYV101-004; 2024-511198-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Refractory Lupus Nephritis; Myasthaenia Gravis; Stiff Person Syndrome; Rheumatoid Arthritis (RA); Multiple Sclerosis; Dermatomyositis; Systemic Sclerosis (SSc)
MeSH Terms: conditions — Lupus Nephritis; Stiff-Person Syndrome; Arthritis, Rheumatoid; Multiple Sclerosis; Dermatomyositis; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: KYV-101

INTERVENTIONS:
Drug: KYV-101 — Autologous fully-human anti-CD19 chimeric antigen receptor T-cell (CD19 CAR T) product.

SUMMARY:
The purpose of this long-term follow-up (LTFU) study is to collect delayed adverse events (AEs) and understand the persistence of KYV-101 (autologous CAR T cell product; gene-modified product), in participants who have been administered KYV-101 (gene-modified product; autologous CAR T cell product).

This LTFU protocol will be open to any participant who received at least one infusion of KYV-101 in a previous Kyverna sponsored clinical trial or Investigator Initiated Trial (IIT).

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent for the LTFU study
* Received at least 1 infusion of KYV-101 as part of a previous KYV-101 parent treatment protocol

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received at least 1 infusion of KYV-101 in a previous KYV-101 treatment clinical study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2041-01 (Estimated); Study Completion 2041-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with new or recurrent malignancies as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with new or exacerbation of a pre-existing neurologic disorder as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with new or exacerbation of a prior rheumatologic or other autoimmune disorder as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with new hematologic disorders as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with new infections as assessed by CTCAE v6.0 through Year 15 of long-term follow-up (LTFU). | Up to 15 years from study entry
Number of participants with positive Replication-Competent Lentivirus (RCL) laboratory test results through Year 5 of long-term follow-up (LTFU). | Up to 5 years from study entry
Number of participants with positive Chimeric Antigen Receptor (CAR) laboratory test results through Year 5 of long-term follow-up (LTFU). | Up to 5 years from study entry
Number of participants with positive Anti-Drug-Antibody (ADA) laboratory test results through Year 5 of long-term follow-up (LTFU). | Up to 5 years from study entry

SECONDARY OUTCOMES:
For lupus nephritis participants, number of participants administered glucocorticoids and other immunosuppressants through Year 2 after KYV101 infusion. | Up to 2 years from first KYV-101 infusion
For stiff-person syndrome participants, change in time required (in seconds) to complete the Timed 25-foot Walk (T25-FW) through Year 4 of LTFU. | Up to 4 years from study entry
  For stiff-person syndrome participants, change in time required (in seconds) from baseline to complete the Timed 25-foot Walk (T25-FW) test as assessed by the investigator through Year 4 of long-term follow-up (LTFU). The T25-FW test is a quantitative mobility and leg function performance test based on a timed 25-foot walk, with shorter times indicating better mobility and improved disease severity.
For myasthenia gravis participants, change in score on the Myasthenia Gravis Activities of Daily Living (MG-ADL) questionnaire through Year 5 of LTFU. | Up to 5 years from study entry
  For myasthenia gravis participants, change in score from baseline on the Myasthenia Gravis Activities of Daily Living (MG-ADL) questionnaire as assessed by the investigator through Year 5 of long-term follow-up (LTFU). The MG-ADL questionnaire is a quantitative functional status instrument, with scores ranging from 0 to 24, with a higher score indicating worse disease severity.
For myasthenia gravis participants, change in score on the Quantitative Myasthenia Gravis (QMG) questionnaire through Year 5 of LTFU. | Up to 5 years from study entry
  For myasthenia gravis participants, change in score from baseline on the Quantitative Myasthenia Gravis (QMG) questionnaire as assessed by the investigator through Year 5 of long-term follow-up (LTFU). The QMG questionnaire is a quantitative muscle strength and endurance/fatigability instrument, with scores ranging from 0 to 39, with a higher score indicating worse disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Denver, Denver, Colorado, United States